CLINICAL TRIAL: NCT01406509
Title: A Phase I Clinical Trial for Safety of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine in Children
Brief Title: Safety of A Group A, C Polysaccharide Meningococcal and Type b Haemophilus Influenzal Conjugate Vaccine in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Royal (Wuxi) Biological Co., LTD (Other)
Responsible Party: Principal Investigator, Fengcai Zhu, Professor, Director of Center for Vaccine Clinical Trials, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT006
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Safety; Conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- children aged 2-5 years (1 dose) (Experimental): group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccines of 0.5ml/dose for a person in 20 children aged 2-5 years, on day 0
  Interventions: Biological: 0.5ml/dose for a person
- children aged 6-23months (2 doses) (Experimental): group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccines of 0.5ml/dose for a person in 20 children aged 6-23 months old, on day 0, 28
  Interventions: Biological: 0.5ml/dose for a person

INTERVENTIONS:
Biological: 0.5ml/dose for a person — group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine of 0.5ml/dose for a person, on day0
  Arms: children aged 2-5 years (1 dose)
Biological: 0.5ml/dose for a person — group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine of 0.5ml/dose for a person, on day0, 28
  Arms: children aged 6-23months (2 doses)

SUMMARY:
Haemophilus influenzae is an important pathogen which can cause primary infection and respiratory viral infection in infants and leaded to secondary infections. The infection of haemophilus is a major cause of morbidity and mortality in infants and children. At present, the developed conjugant Hib vaccine is proved to be safe and effective, 90-99% of children will produce antibody of protection after 3 doses. Because Hib vaccine can prevent meningitis, pneumonia, epiglottis inflammation and other serious infection caused by Hib bacteria, the WHO suggested that Hib vaccine should be included in the infant's normal immune programming.

Since the use of meningitis aureus polysaccharide vaccine, incidence of a disease in recent years is declined and maintain to the level of 0.5 per 1/100 thousand. But meningitis aureus polysaccharide vaccine with a relatively poor immune response in the infants under the age of two, and the remaining 60% with a low antibody level and a short duration.

According to the present immunization schedule, to reach the median level of antibody levels there are at least 4 doses in need. So it is meaningful to improving vaccine immunogenicity, to provide high levels of long-term protection and to reduce the number of injections.

The objective of this study is to evaluate the safety of the group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged from 6 months to 5years old of normal intelligence
* The subjects'guardians are able to understand and sign the informed consent
* Subjects established as healthy after medical history questioning,physical examination and clinical decision and in accordance with vaccination requirements of the experimental vaccine
* Subjects who can comply with the requirements of the clinical trial program according to the researcher's views
* Subjects who have never received group A, C polysaccharide meningococcal vaccine and type b haemophilus Influenzal vaccine
* Subjects with temperature <37°C on axillary setting

Exclusion Criteria:

Exclusion Criteria for the first dose:

* Subject who has a medical history of Meningitis
* Subject that has a medical history of any of the following: allergies, seizures, epilepsy, encephalopathy history and so on
* Subject who is allergic with tetanus toxoid components
* Subject suffering from thrombocytopenia or other coagulation disorder may lead to contraindication to intramuscular injection
* Subject who has a history of allergic reactions
* Any known immunological dysfunction
* Had received gamma globulin or immune globulin, in the past two weeks
* Subject suffering from congenital malformations, dysgenopathy or serious chronic disease
* Any acute infections
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion Criteria for the second dose:

* Had any Grade 3 or Grade 4 adverse reactions or events
* Any situation meets the exclusion criteria stated in the exclusion criteria for first dose
* Any condition the investigator believed may affect the evaluation of the vaccine

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The adverse reactions in healthy children (2-5 years) after the first vaccination | 7 days after the first vaccination
  to evaluate the adverse reactions of the group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine in healthy children (2-5 years) after the first vaccination
The adverse reactions in healthy children (6-23 months) after the first vaccination | 7 days after the first vaccination
  to evaluate the adverse reactions of the group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine in healthy children (6-23 months) after the first vaccination
The adverse reactions in healthy children (6-23 months) after the second vaccination | 7 days after the second vaccination
  to evaluate the adverse reactions of the group A, C polysaccharide meningococcal and type b haemophilus Influenzal Conjugate vaccine in healthy children (6-23 months) after the second vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China